CLINICAL TRIAL: NCT03869788
Title: Parasitological Evaluation of Fascioliasis in Clinically Suspected Patients and the Effect of Some Plant Extract on The Adult Worm
Brief Title: Parasitological Evaluation of Fascioliasis in Clinically Suspected Patients .
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Samah Mohammad Hussein, Teaching assistant at parasitology department, Assiut University
Other Study IDs: PEOFCSP
Record Dates: First submitted 2019-03-06; First posted 2019-03-11 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-03

CONDITIONS: Fascioliasis
MeSH Terms: conditions — Fascioliasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — Stool samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
WHO considers foodborne trematodes as neglected tropical diseases. Fascioliasis is the most widely distributed trematode reported from over 81 countries around the world it imposes its highest burden in developing countries

DETAILED DESCRIPTION:
liver flukes are disease affecting herbivorous animals and caused by Fasciola hepatica and Fasciola gigantica In Egypt, donkeys and camels as well, are hosts for Fasciola gigantica. Fascioliasis also affects man . number of humans infected with Fasciola spp. has been estimated at 2.6 million . Globally, fascioliasis due to both fluke species is conservatively thought to cause production losses of over US$3 billion per annum .

These infection sources include foods, water and combinations of both. Ingestion of freshwater wild plants is the main source, with watercress and secondarily other vegetables involved. . Drinking of contaminated water, beverages and juices, ingestion of dishes and soups and washing of vegetables, fruits, tubercles and kitchen utensils with contaminated water are increasingly involved .

. Two clinical stages are recognized in humam fascioliasis: An acute stage coincides with the larval migration and worm maturation in the hepatic tissue, and a chronic stage coincides with the persistence of Fasciola worms in the bile ducts

* the acute phase of fascioliasis is characterized by fever, abdominal pain, hepatosplenomegaly, gastrointestinal disturbances, skin rashes, high leukocyte count, eosinophilia, anemia, and elevated erythrocyte sedimentation rate (ESR); abnormal liver function tests have also been reported .
* The latent phase is characterized by nonspecific symptoms, including vague gastrointestinal disturbances, and intermittent eosinophilia.
* The chronic phase is characterized by regular and constant biliary obstruction; symptoms include biliary colic pain, intermittent jaundice, eosinophilia, and right upper-quadrant abdominal tenderness. However, the percentage of asymptomatic infections is high .

Triclabendazole (TCBZ) is a benzimidazole derivative and is the current drug of choice for treating fascioliasis. What sets TCBZ aside from the other available fasciolicides is its ability to target flukes from as early as 3 days old right through to the fully mature stages ,. Due to the high prevalence of TCBZ resistance (TCBZ-R), effective management of drug resistance is now critical for sustainable livestock production Wich highlights the importance of plant essential oils as novel anti-parasitic agents; Some plant oils have immunomodulatory effects that could modify host- parasite immunobiology In addition, the safety and use of plant essential oils in drug resistant cases are considered the most advantages.

Allium sativum commonly called garlic belongs to the family Alliaceae. It has been used for centuries to fight infections as an antioxidant ,antibacterial, antiviral, antifungal , anti-parasitic , antihypertensive , anthelmintic, and anti- diabetic agent .

Lately, the anthelmintic effect of garlic has been a matter of interest of researchers .

It's Potentially Active Chemical Constituents are :

* Sulfur compounds: aliin, allicin, ajoene, allylpropyl disulfide, diallyl trisulfide, s- allylcysteine, vinyldithiines, S-allylmercaptocystein, and others .
* Enzymes: allinase, peroxidases, myrosinase, and others .
* Amino acids and their glycosides: arginine and others .
* Selenium, germanium, tellurium and other trace minerals . Cloves (Syzygium aromaticum) Are the dried flower buds of an aromatic tree that is used as a spice. It mainly contains volatile oil, i.e. eugenol 81.1%, caryophyllin, tannins and gum.Clove oil has been used as analgesic, antibacterial, anticonvulsant, anticoagulant, antifungal, anti-inflammatory, antioxidant, antiseptic, antitumor, antiviral, disinfectant, immune stimulant as well as insecticidal .

Nanotechnology has a wide range of action in sciences like medicine, electronics, food and agriculture. Its application has strengthen systems to control diseases in animals, water disinfection, safety in systems of food supply, energy conversion, plague localization technology, advances in fast detection of morphological changes in the physicochemical properties of food, increment in nutrient value, quality control, food security, development of novel products and packing design .

It is the current trend in research field, using small size of materials with wide range of application . In nanotechnology there is treatment of atom, molecules or compounds to produce nanoparticle with different properties .The size and structure of nanoparticle is similar to most biological molecules, therefore nano particle can be useful for in research .

There are many types of nanoparticles: organic, inorganic, nanocrystals, nanotubes, polymeric structures such as dendrimers, etc. They are used primarily in research and drug delivery systems .

In that research garlic and cloves will be used in vitro to detect their fasciolicidal effects on adult Worm obtained from locally slaughtered animals .

ELIGIBILITY:
Inclusion Criteria:

* vague gastrointestinal disturbances.
* intermittent eosinophilia.
* biliary obstruction.
* biliary colic pain.
* intermittent jaundice.
* right upper-quadrant abdominal tenderness.

Exclusion Criteria:

* no exclusion Criteria

Ages: 16 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: * Human cases complaining of previous symptoms .
  * Farmer .
  * Resident of rural area in Assiut governorate especially in Manfalout city .
  * Exposed to stagnant chanell water .
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2020-03-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
Number of human cases whose stool examination positive for fasciola eggs . | One year
  Stool analysis will be done to detect eggs of fasciola worm by direct smear and concentration techniques .
  to patients complaining of vague gastrointestinal disturbances, and biliary colic pain, intermittent jaundice and right upper quadrant abdominal tenderness .

CONTACTS AND LOCATIONS:
Overall Officials: Salma M Abdel-Rahman, prof, Study Director — unaffiliation
Locations (1):
- Assiut University Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Nahed HA, Hoda AT, Yomna IM. Effects of garlic on albino mice experimentally infected with Schistosoma mansoni: a parasitological and ultrastructural study. Trop Biomed. 2009 Apr;26(1):40-50. PMID 19696726